CLINICAL TRIAL: NCT07195864
Title: Retrospective Chart Review of Patients With Acanthamoeba Keratitis Who Have Received 0.8 mg/mL Polihexanide as Part of the "Medicines in Special Situations" (Medicamentos en Situaciones Especiales) Program in Spain.
Status: Recruiting | Type: Observational
Sponsor: SIFI SpA (Industry)
Responsible Party: Sponsor
Other Study IDs: 059/SI
Record Dates: First submitted 2025-09-02; First posted 2025-09-29 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Acanthamoeba Keratitis
Keywords: Acanthamoeba Keratitis PHMB
MeSH Terms: conditions — Acanthamoeba Keratitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: PHMB 0.08% — The study population for this study is patients diagnosed with AK treated with 0.8 mg/ml polihexanide as part of the Spanish Medicines in Special Situations program.

SUMMARY:
The study will be a multicentric, retrospective, non-interventional medical chart review of patients with AK who initiated a treatment with 0.8 mg/ml polihexanide as part of the Spanish Medicines in Special Situations program, whether they fully completed the treatment or not.

Baseline date is defined as the date of 0.8 mg/ml polihexanide initiation. The Study Period for each patient will be considered the period from the baseline to the conclusion of the treatment.

DETAILED DESCRIPTION:
Primary objective:

• To describe the efficacy of 0.8 mg/ml polihexanide in the clinical resolution of AK in all patients that satisfy the inclusion criteria of the study, as measured by the proportion of patients cured at the end of the study period, confirmed at the 30-day follow-up (when available).

Secondary objectives:

• To describe the efficacy of 0.8 mg/ml polihexanide in the clinical resolution of AK in full compliant patients.

• To describe the efficacy of 0.8 mg/ml polihexanide in the improvement of visual acuity (VA).

• To describe the efficacy of 0.8 mg/ml polihexanide in the improvement of ocular clinical findings.

• To describe de efficacy of 0.8 mg/ml polihexanide in the reduction of pain.

• To determine the rate of patients requiring ocular surgery.

• To determine the rate of patients using topical ophthalmologic steroids or other relevant medications.

• To determine the time from start of treatment until clinical resolution.

• To determine the proportion of patients with concomitant fungal or bacterial corneal infections.

• To describe the efficacy of 0.8 mg/ml polihexanide in preventing disease relapse.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the Spanish Medicines in Special Situations (Gestión de Medicamentos en Situaciones Especiales) program from August 2022 to 31 October 2024, because they presented clinical signs and symptoms consistent with AK and the identification of Acanthamoeba was confirmed by at least one of the following techniques:

o Confocal Microscopy o PCR o Identification by microbiological culture or cytological smear.

• Diagnosis of AK at least 2 months before inclusion in the study

• Age ≥12 years at the time of diagnosis.

• To have started and completed the treatment with 0.8 mg/ml polihexanide at the moment of the inclusion.

Exclusion Criteria:

* No participation in another trial contemporary at this one

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population for this study is patients diagnosed with AK treated with 0.8 mg/ml polihexanide as part of the Spanish Medicines in Special Situations program.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
the proportion of patients cured at the end of the study period, confirmed at the 30-day follow-up (when available) | The end of the study period, confirmed at the 30-day follow-up (when available).
  The primary endpoint will be the proportion of patients cured at the end of the study period, confirmed at the 30-day follow-up (when available). The primary analysis will be performed on all patients that satisfy the inclusion criteria of the study
The primary endpoint will be the proportion of patients cured at the end of the study period, confirmed at the 30-day follow-up (when available). | he end of the study period, confirmed at the 30-day follow-up (when available).
  The primary endpoint will be the proportion of patients cured at the end of the study period, confirmed at the 30-day follow-up (when available). The primary analysis will be performed on all patients that satisfy the inclusion criteria of the study.

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - HU Ramon y Cajal, Madrid, Principality of Asturias
  - HU La Paz, Madrid
  - IO Fernandez Vega, Madrid
  - CHUO Ourense, Ourense

IPD SHARING:
Plan to Share IPD: No